CLINICAL TRIAL: NCT04868149
Title: Clinical Outcome and Future Liver Remnant Regenerative Response in Laparoscopic Versus Open ALPPS: A Randomized Clinical Trial
Brief Title: Clinical Outcome and Future Liver Remnant Regenerative Response in Laparoscopic Versus Open ALPPS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Albert Chi Yan Chan, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UW20-599
Record Dates: First submitted 2020-12-28; First posted 2021-04-30 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Liver Cancer
Keywords: ALPPS; Small future liver remnant; Liver cancer; Hepatocellular carcinoma; Liver metastasis; Laparoscopic surgery; Minimal invasive
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patient are randomly assigned into either open or laparoscopic approach. The ratio of open and laparoscopic is 1:1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic ALPPS (Experimental): Laparoscopic ALPPS procedure
  Interventions: Procedure: Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS)
- Open ALPPS (Active Comparator): Open ALPPS procedure
  Interventions: Procedure: Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS)

INTERVENTIONS:
Procedure: Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) — Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) is a surgical procedure that induces rapid liver regeneration in patients with small liver remnant planning for major liver resection. It is a two-staged operation with stage I including portal vein ligation and splitting the right liver away from the left liver. After stage I, the left liver will undergo rapid liver regeneration and the stage II operation can be performed at 7-10 days after stage I operation when the liver remnant reaches an adequate size. In stage II operation, the right liver that contains the tumor is then removed.
  Other Names: ALPPS

SUMMARY:
Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) is a new surgical procedure that induces rapid liver regeneration in patients with small liver remnant planning for major liver resection. It is a two-staged operation with stage I including portal vein ligation and splitting the right liver away from the left liver. After stage I, the left liver will undergo rapid liver regeneration and the stage II operation can be performed at 7-10 days after stage I operation when the liver remnant reaches an adequate size. In stage II operation, the right liver that contains the tumor is then removed. This surgical procedure was incepted in Germany in 2013 and was later started in Queen Mary Hospital in Hong Kong for the first time in December 2015. The initial indication was mainly for colorectal liver metastasis but due to the relatively high incidence of hepatocellular carcinoma in Hong Kong, HBP surgery team of Queen Mary Hospital has transferred this procedure to be applied for hepatitis-related hepatocellular carcinoma and so far, the centre has cumulated one of the largest single-center experience in the literature. Nonetheless, the usual approach for ALPPS involved open surgery and induced substantial surgical stress to the patient, especially after stage I operation. With the advent of minimally invasive liver surgery in recent years, the team has successfully applied laparoscopic surgery to ALPPS in 2019. Despite the advancement in laparoscopic surgical skills that rendered laparoscopic ALPPS feasible, there is scarcity of data in the literature to evaluate its outcome in comparison with open ALPPS with regard to perioperative recovery and liver regeneration. Hence, the aim of this project is to evaluate the short-term clinical outcomes of laparoscopic ALPPS and the impact of laparoscopy on liver remnant regeneration after ALPPS in a prospective randomised clinical trial setting.

DETAILED DESCRIPTION:
Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) has been popularized as an alternative approach for FLR augmentation in recent years. The main indication at the early phase of development of this procedure was bilobar colorectal liver metastasis, or other non-primary liver tumors. Since 2015, HBP surgery team of Queen Mary Hospital has started to transfer this novel approach to treat patients with hepatitis-related hepatocellular carcinoma and small future liver remnant contemplating for major hepatectomy. Despite the initial global enthusiasm to embark on ALPPS, the procedure was criticized for its high postoperative morbidity and mortality rates. However, through the establishment of the international ALPPS registry and familiarization of the procedure, the outcome of ALPPS has been benchmarked and standardized with a mortality rate <4%. The initial experience of ALPPS for HCC was also reported. With cumulative experience, ALPPS has become a safe and effective treatment approach for surgical modulation of insufficient FLR when compared with the conventional approach in the form of portal vein embolization. Nonetheless, ALPPS is a two-stage procedure that commonly involved an open laparotomy. However, the postoperative pain control and speed of recovery after stage I ALPPS would be affected by the substantial surgical stress induced by laparotomy. On the other hand, the rapid development of laparoscopic surgery has rendered laparoscopic liver surgery a much more feasible and safer surgical approach in recent years. As such, minimally invasive approach becomes an attractive option for ALPPS, at least for stage I procedure. Data on the application of laparoscopic ALPPS remained scarce with only one study reported the short-term outcome in a series of 10 patients predominantly affected by colorectal liver metastasis.

Since the short-term postoperative safety profile and underlying intraoperative haemodynamic changes induced by ALPPS for hepatitis-related HCC under conventional open approach was ascertained by our recent study, it is considered that it is the right time to introduce laparoscopy for ALPPS and to compare its clinical outcome with open approach. To date, a total of 4 patients have received laparoscopic ALPPS in the centre.

Recent studies suggested that laparoscopic liver resection may be associated with reduced inflammatory and stress response as compared with open resection as indicated by a reduced expression of inflammatory cytokines such as interleukin-6, tumor necrosis factor. On the other hand, study on liver regeneration after open ALPPS showed an elevated gene expression of IL-6 and TNF as well as increased plasma levels within 24 hours after the procedure when compared with portal vein ligation. It remains uncertain if reduced level of cytokines or inflammatory markers induced by laparoscopy would affect the liver regeneration rate in ALPPS patients and its clinical outcome. Hence, there is a need to clarify this issue in the current project.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of malignant liver tumor contemplating for extended right hepatectomy or right trisectionectomy
2. Patient consent
3. Age >/= 18
4. FLR/ESLV </= 30%
5. Indocyanine green clearance rate at 15 mins : < 18%
6. Platelet count > 100x10^9/L
7. Child A cirrhosis (due to hepatitis B/C virus, or alcohol, or autoimmune disease)
8. American Society of Anaesthesiology score < 3
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Technical factors eligible for laparoscopic ALPPS

* single long-segment portal

Exclusion Criteria:

1. Absence of consent
2. Decompensated liver disease as indicated by the presence of ascites, varices and hepatic encephalopathy
3. ECOG performance status >/= 3
4. Main portal vein thrombosis
5. FLR/ESLV > 30%

Technical factors not eligible for laparoscopic ALPPS

* Short-segment right portal vein or early bifurcation of right anterior/posterior portal vein, or other portal vein anomalies
* Large tumor size with diameter > 5 cm
* Intolerance to CO2 pneumoperitoneum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of future liver remnant volume increment by percentage after stage I ALPPS | During hospital stay after stage I ALPPS, an average of 1-2 weeks
  Amount of future liver remnant volume increment by percentage after stage I ALPPS

SECONDARY OUTCOMES:
Preoperative blood loss during stage 1 ALPPS | During hospital stay after stage I ALPPS, an average of 1-2 weeks
  Preoperative blood loss during stage 1 ALPPS
Length of hospital stay after stage 1 ALPPS | During hospital stay after stage I ALPPS, an average of 1-2 weeks
  Length of hospital stay after stage 1 ALPPS
Overall morbidity in number and mortality rates in percentage after stage 1 ALPPS | During hospital stay after stage I ALPPS, an average of 1-2 weeks
  Overall morbidity and mortality rates after stage 1 ALPPS
Inflammatory markers associated with inflammation and regeneration after stage 1 ALPPS | During hospital stay after stage I ALPPS, an average of 1-2 weeks
  Inflammatory markers e.g. IL-6 (pg/ml), IL-8 (pg/ml) and TNF-alpha (pg/ml) associated with inflammation and regeneration after stage 1 ALPPS

CONTACTS AND LOCATIONS:
Overall Officials: Albert Chan, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang H, de Santibanes E, Schlitt HJ, Malago M, van Gulik T, Machado MA, Jovine E, Heinrich S, Ettorre GM, Chan A, Hernandez-Alejandro R, Robles Campos R, Sandstrom P, Linecker M, Clavien PA. 10th Anniversary of ALPPS-Lessons Learned and quo Vadis. Ann Surg. 2019 Jan;269(1):114-119. doi: 10.1097/SLA.0000000000002797. PMID 29727331
- [Result] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038
- [Result] Schadde E, Ardiles V, Robles-Campos R, Malago M, Machado M, Hernandez-Alejandro R, Soubrane O, Schnitzbauer AA, Raptis D, Tschuor C, Petrowsky H, De Santibanes E, Clavien PA; ALPPS Registry Group. Early survival and safety of ALPPS: first report of the International ALPPS Registry. Ann Surg. 2014 Nov;260(5):829-36; discussion 836-8. doi: 10.1097/SLA.0000000000000947. PMID 25379854
- [Result] Linecker M, Bjornsson B, Stavrou GA, Oldhafer KJ, Lurje G, Neumann U, Adam R, Pruvot FR, Topp SA, Li J, Capobianco I, Nadalin S, Machado MA, Voskanyan S, Balci D, Hernandez-Alejandro R, Alvarez FA, De Santibanes E, Robles-Campos R, Malago M, de Oliveira ML, Lesurtel M, Clavien PA, Petrowsky H. Risk Adjustment in ALPPS Is Associated With a Dramatic Decrease in Early Mortality and Morbidity. Ann Surg. 2017 Nov;266(5):779-786. doi: 10.1097/SLA.0000000000002446. PMID 28806301
- [Result] Chan AC, Pang R, Poon RT. Simplifying the ALPPS procedure by the anterior approach. Ann Surg. 2014 Aug;260(2):e3. doi: 10.1097/SLA.0000000000000736. No abstract available. PMID 24866543
- [Result] Chan AC, Poon RT, Chan C, Lo CM. Safety of ALPPS Procedure by the Anterior Approach for Hepatocellular Carcinoma. Ann Surg. 2016 Feb;263(2):e14-6. doi: 10.1097/SLA.0000000000001272. No abstract available. PMID 26079914
- [Result] Raptis DA, Linecker M, Kambakamba P, Tschuor C, Muller PC, Hadjittofi C, Stavrou GA, Fard-Aghaie MH, Tun-Abraham M, Ardiles V, Malago M, Campos RR, Oldhafer KJ, Hernandez-Alejandro R, de Santibanes E, Machado MA, Petrowsky H, Clavien PA. Defining Benchmark Outcomes for ALPPS. Ann Surg. 2019 Nov;270(5):835-841. doi: 10.1097/SLA.0000000000003539. PMID 31592812
- [Result] Chan A, Zhang WY, Chok K, Dai J, Ji R, Kwan C, Man N, Poon R, Lo CM. ALPPS Versus Portal Vein Embolization for Hepatitis-related Hepatocellular Carcinoma: A Changing Paradigm in Modulation of Future Liver Remnant Before Major Hepatectomy. Ann Surg. 2021 May 1;273(5):957-965. doi: 10.1097/SLA.0000000000003433. PMID 31305284
- [Result] Machado MA, Makdissi FF, Surjan RC, Basseres T, Schadde E. Transition from open to laparoscopic ALPPS for patients with very small FLR: the initial experience. HPB (Oxford). 2017 Jan;19(1):59-66. doi: 10.1016/j.hpb.2016.10.004. Epub 2016 Nov 2. PMID 27816312
- [Result] Burpee SE, Kurian M, Murakame Y, Benevides S, Gagner M. The metabolic and immune response to laparoscopic versus open liver resection. Surg Endosc. 2002 Jun;16(6):899-904. doi: 10.1007/s00464-001-8122-x. Epub 2002 Feb 27. PMID 12163951
- [Result] Schlegel A, Lesurtel M, Melloul E, Limani P, Tschuor C, Graf R, Humar B, Clavien PA. ALPPS: from human to mice highlighting accelerated and novel mechanisms of liver regeneration. Ann Surg. 2014 Nov;260(5):839-46; discussion 846-7. doi: 10.1097/SLA.0000000000000949. PMID 25379855